CLINICAL TRIAL: NCT01958567
Title: Optical Coherence Tomography in the Diagnosis of Scleritis and Episcleritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Eye Center and The Eye Foundation for Research in Ophthalmology (Other)
Responsible Party: Principal Investigator, Samir S. Shoughy, MD, FRCS (Glasg.), Ophthalmologist, The Eye Center and The Eye Foundation for Research in Ophthalmology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TEC 125; TEC 2013-006 [THE EYE CENTER]
Record Dates: First submitted 2013-10-07; First posted 2013-10-09 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Scleritis and Episcleritis
Keywords: Scleritis; Episcleritis; Optical coherence Tomography
MeSH Terms: conditions — Scleritis | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with clinical signs of scleritis or episcleritis (Experimental): Optical Coherence Tomography for patients with scleral inflammation
  Interventions: Other: Optical Coherence Tomography
- Normal subjects with normal sclera (Experimental): Optical Coherence Tomography on eyes with normal scleral
  Interventions: Other: Optical Coherence Tomography

INTERVENTIONS:
Other: Optical Coherence Tomography

SUMMARY:
The main purpose of this study is to describe the optical coherence tomography (OCT) findings in eyes with scleral inflammation and to differentiate cases with anterior scleritis from those with episcleritis and normal controls.

DETAILED DESCRIPTION:
A total of 40 eyes will be included. 20 eyes with scleral inflammation and 20 eyes from healthy subjects as controls. Each patient will undergo complete ophthalmic and medical examination. Laboratory studies will performed whenever indicated. Optical coherence tomography B-scans of the sclera in the perilimbal area will done for all cases.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 years any gender
* Patients with clinical signs of scleritis or episcleritis
* Signed informed consent

Exclusion Criteria:

* Infectious keratitis or conjunctivitis
* Patients 18 years or younger
* Inability to open the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-07; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To describe the optical coherence tomography (OCT) findings in eyes with scleral inflammation | 3 months
  To differentiate cases with anterior scleritis from those with episcleritis and normal controls

CONTACTS AND LOCATIONS:
Locations (1):
- The Eye Center, Riyadh, Saudi Arabia